CLINICAL TRIAL: NCT05356091
Title: Comparison of Postoperative Recovery Quality Between Sevoflurane and Remimazolam for General Anesthesia for Transurethral Resection of Bladder Tumor
Brief Title: Quality of Recovery of Remimazolam Versus Sevoflurane in Transurethral Bladder Resection.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kangbuk Samsung Hospital (Other)
Collaborators: Hana Pharm Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Eunah Cho, MD, Assistant Professor, Kangbuk Samsung Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: QRST
Record Dates: First submitted 2022-04-24; First posted 2022-05-02 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Quality of Recovery
MeSH Terms: interventions — Sevoflurane; remimazolam

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sevoflurane (Active Comparator): General anesthesia using sevoflurane
  Interventions: Drug: Sevoflurane
- Remimazolam (Experimental): General anesthesia using remimazolam
  Interventions: Drug: Remimazolam

INTERVENTIONS:
Drug: Sevoflurane — Sevoflurane is chosen as an anesthetic agent for general anesthesia. General anesthesia for the patients in this group will be induced with propofol (1-1.5 mg/kg), and will be maintained with sevoflurane to keep patient state index of 25-50.
  Arms: Sevoflurane
Drug: Remimazolam — Remimazolam is chosen as an anesthetic agent for general anesthesia. General anesthesia for the patients in this group will be induced with remimazolam, and will be maintained with remimazolam to keep patient state index of 25-50.
  Arms: Remimazolam

SUMMARY:
This study was designated to investigate the quality of recovery after transurethral bladder resection. Because, patients undergoing transurethral bladder resection are mostly old age, and because of catheter-related bladder discomfort are common after transurethral bladder resection, study on the quality of recovery after transurethral bladder resection seems to be meaningful. In general, sevoflurane is commonly used as an anesthetic agent for general anesthesia of transurethral bladder resection. The purpose of this study is to investigate whether remimazolam is not inferior to sevoflurnane in terms of quality of recovery after transurethral bladder resection.

ELIGIBILITY:
Inclusion Criteria:

* adult patients aged from 19 years
* Americaln Society of Anesthesiologist's class I, II, and III
* scheduled to undergo elective transurethral bladder resection under general anesthesia

Exclusion Criteria:

* refuse to participate in the study
* cannot read, or sign the consent form (e.g., iliterate, foreigner, eye disease)
* history of allergy to benzodiazepines
* decreased liver, kidney, or heart function
* pregnant women or breastfeeding patients
* history of drug or alcohol abuse
* obesity (body mass index > 30kg/m2)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2022-12-02 (Actual); Primary Completion 2023-02-24 (Actual); Study Completion 2023-02-24 (Actual)

PRIMARY OUTCOMES:
Quality of recovery -15 score at postoperative day 1 | postoperative day 1
  Quality of recovery-15 questionnaire, which consists 15 questions. The score ranges from 0 to 150. The higher the score, the better the quality of recovery.

SECONDARY OUTCOMES:
Catheter related bladder discomfort | 5 minutes, and 1 hour after post-anesthesia circuit unit arrival.
  Catheter related bladder discomfort is assessed as none, mild, moderate and severe.

CONTACTS AND LOCATIONS:
Overall Officials: Eunah Cho, Pf., Principal Investigator — KangbukSamsung Hospital
Locations (1):
- Eunah Cho, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided